CLINICAL TRIAL: NCT04799639
Title: Efficacy and Toxicity of Paclitaxel, Cisplatin Combined With Sindilimab in Neoadjuvant Chemotherapy for Locally Advanced Cervical Cancer
Brief Title: Efficacy and Toxicity of Paclitaxel, Cisplatin Combined With Sindilimab in NACT for Locally Advanced Cervical Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jihong Liu, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2020-201-01
Record Dates: First submitted 2021-03-14; First posted 2021-03-16 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Cervical Cancer; Chemotherapy Effect; Programmed Cell Death 1 Receptor / Antagonists & Inhibitors; Neoadjuvant Therapy
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: patients will receive intravenous drip of standard dose paclitaxel + cisplantin + Sindilimab every 3 weeks for 3 cycles
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- paclitaxel + cisplantin + Sindilimab (Experimental): standard dose paclitaxel + cisplantin + Sindilimab every 3 weeks for 3 cycles paclitaxel 150mg/m2，ivdrip,>3 hours cisplantin 70mg/m2，ivdrip，>1 hours Sindilimab 200mg，ivdrip, >0.5 hours
  Interventions: Drug: Sindilimab +paclitaxel+ cisplantin

INTERVENTIONS:
Drug: Sindilimab +paclitaxel+ cisplantin — standard dose paclitaxel + cisplantin + Sindilimab every 3 weeks for 3 cycles

SUMMARY:
To determine the safety and efficacy of Sindilimab combined with Paclitaxel and Cisplatin in neoadjuvant chemotherapy for Locally Advanced Cervical Cancer

DETAILED DESCRIPTION:
A total of 47 patients will be enrolled in this study. After screening, patients will receive intravenous drip of standard dose paclitaxel + cisplantin + Sindilimab every 3 weeks for 3 cycles. CT/MR of chest, upper and lower abdomen and pelvic MR will be performed before treatment and 2 weeks after the 3rd cycle chemotherapy. The objective response rate (ORR) (CR + PR) is evaluated by comparing with baseline based on RECISTv1.1. Radical surgery will be performed after NACT. According to the postoperative pathological results, the pathological complete remission rate (pCR) will be evaluated. The adverse events will be continuously monitored during treatment until 30 days after chemotherapy. Toxic adverse events is evaluated according to NCI-CTCAEv5.0 criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 to 65 years with primary cervical cancer;
2. Clinical diagnosis of cervical cancer stage IB3 or IIA2 (FIGO stage, 2018). The stage was determined by two associate senior physicians or above after examining the patients;
3. no distant organ metastasis, and the short diameter of retroperitoneal lymph nodes was less than 1 cm;
4. according to the RECIST version 1.1 criteria, the measurable lesion of the cervix assessed by imaging was > 3.5 cm;
5. histological types includes cervical squamous cell carcinoma, adenocarcinoma or adenosquamous carcinoma;
6. no radiotherapy, chemotherapy or targeted therapy before;
7. the expected survival time was greater than 3 months;
8. the ECOG score of the Eastern Cooperative Oncology Group was 0 - 1;
9. the function of important organs met the requirements of surgery, chemotherapy and radiotherapy.

Exclusion Criteria:

1. Patients with other malignant tumors;
2. Patients is pregnancy or in perinatal period;
3. Patients with myocardial infarction or stroke, or unstable angina pectoris, decompensated heart failure, or deep venous thrombosis;
4. Patients with NCI-CTCAE 5.0 ≥ grade 2 arrhythmia, any grade of atrial fibrillation, or clinically significant supraventricular or ventricular arrhythmia requiring treatment or intervention;
5. Patients with active pneumonia: hepatitis patients with progressive loss of appetite, general weakness, nausea, acid reflux, anorexia, abdominal distension and other clinical manifestations, abnormal liver function and jaundice such as yellow eyes, yellow urine and other clinical symptoms;
6. Patients with liver dysfunction (aspartate/alanine aminotransferase > 2.5 times the upper limit of the standard);
7. Patients with renal insufficiency (serum creatinine > 2 times the upper limit of the standard);
8. History of chronic lung disease with restrictive respiratory dysfunction;
9. History of important organ transplantation, history of immune diseases;
10. History of severe mental illness, History of cerebral dysfunction;
11. history of drug abuse or drug use;
12. patients are using immunosuppressive agents, or systemic hormone therapy to achieve the purpose of immunosuppression (dose > 10 mg prednisone or other effective hormones), and continue to use 2 weeks before enrollment;
13. coagulation abnormalities (INR > 2.0, PT > 16s), with bleeding tendency or are receiving thrombolytic or anticoagulant therapy, allowing prophylactic use of low-dose aspirin,Low molecular weight heparin;
14. Congenital or acquired immunodeficiency (such as HIV infection);
15. Received live vaccine within 30 days before the first dose;
16. Unable or unwilling to sign the informed consent form or comply with the study requirements;
17. Have a history, disease or laboratory abnormalities that may interfere with the test results or prevent the subject from participating in the study, or the investigator believes that participating in the study is not in the best benefit of the subject.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2021-03-18 (Actual); Primary Completion 2024-06-17 (Actual); Study Completion 2024-06-24 (Actual)

PRIMARY OUTCOMES:
pathological complete remission rate (pCR) rate | 3 months
  According to the postoperative pathological results, the pathological complete remission rate (pCR) will be evaluated.

SECONDARY OUTCOMES:
objective response rate (ORR) (CR + PR) | 3 months
  The objective response rate (ORR) (CR + PR) is evaluated by comparing with baseline based on RECISTv1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Jihong Liu, Ph.D., Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University cancer center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No